CLINICAL TRIAL: NCT06921031
Title: Stroke Patients' Preferences for an Exoskeleton for Lower Limb Rehabilitation Using the DCE Method.
Brief Title: Stroke Patients' Preferences for an Exoskeleton for Lower Limb Rehabilitation Using the DCE Method (EXOPREF)
Acronym: EXOPREF
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0363 - EXOPREF
Record Dates: First submitted 2025-03-17; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: Chronic Stroke Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of this study is to investigate the preferences of individual stroke patients for key features of an exoskeleton, intended for lower limb rehabilitation, with a view to its potential integration into the design of future exoskeletons. This will be a multicenter study. Patients will be presented different scenarios of choices about the attributes about gait exoskeleton.

Conditional logistic regression models will be used to define the preferences of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* informed consent to participate in the study
* motor impairment secondary to stroke
* ability to answer the questionnaire with or without assistance from a relative or interviewer

Exclusion Criteria:

- history of lower-limb exoskeleton use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic stroke patients without any specific characteristics
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Choices of the participants | One hour
  The study will describe the distribution of participants' choices among the scenarios presented in the experiment.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Brest, Brest
  - Centre de rééducation Kerpape, Ploemeur

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement